CLINICAL TRIAL: NCT01490983
Title: Pilot Study to Assess Telemonitoring of Gleevec (Imatinib Mesylate) or Tasigna (Nilotinib) Therapy
Brief Title: Telemonitoring Study - for Chronic Myeloid Leukemia (CML)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to lack of funding
Sponsor: Rex Cancer Center, Raleigh, NC (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Leap of Faith Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: RexCCWF1
Record Dates: First submitted 2011-12-08; First posted 2011-12-13 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2016-04

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic Myeloid Leukemia; Chronic Phase CML
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- eMedonline access (Experimental): patients will have access to eMedonline access for 3 months
  Interventions: Behavioral: eMedonline access
- no access to eMedonline (Other): patients will be followed for 3 months with no access to eMedonline
  Interventions: Behavioral: no access to eMedonline

INTERVENTIONS:
Behavioral: no access to eMedonline — patients will be followed for 3 months but will not use eMedonline
  Other Names: Telemonitoring system; e-diary; electronic diary
  Arms: no access to eMedonline
Behavioral: eMedonline access — patients will be given access to eMedonline use for 3 months
  Other Names: Telemonitoring system; e-diary; electronic diary
  Arms: eMedonline access

SUMMARY:
This study is being conducted in a population of patients with chronic phase Chronic Myeloid Leukemia (CML) to learn more about how patients follow prescribed regimens for taking oral cancer drugs.

DETAILED DESCRIPTION:
This is a randomized, controlled pilot study to introduce eMedonline telemonitoring technology to CML patients taking Gleevec or Tasigna. eMedonline will be used to automatically collect time-dose specific medication data for individual patients, including dosing times, missed doses, adverse events and e-diary data. All data will be available to research staff for remote review via Web interface. Adverse events and non-adherence will prompt interventions including supportive care counseling.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older.
* Pathologically documented diagnosis of Chronic Phase CML (Ph+) in whom treating physician has determined that treatment with imatinib or nilotinib is appropriate
* Patients currently receiving Gleevec (imatinib) 300-600 mg daily or Tasigna (nilotinib) 300-400 mg twice daily
* ECOG Performance status 0, 1, or 2
* Adequate end organ function, defined as:

  * Total bilirubin < 1.5 xULN
  * SGOT and SGPT <2.5 x ULN
  * Creatinine < 1.5 x ULN
  * ANC > 1.5
  * Platelets > 100,000
* Female patients of child bearing potential must have a negative urine or serum pregnancy test at screening.
* Patient is able to read and speak English
* Patient is willing and able to use a cell phone
* Written, voluntary informed consent

Exclusion Criteria:

* Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-04; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
eMedonline will be used to measure non-compliance in taking oral drug regimens. | at 6 months, non-compliance will be measured in each arm of study
  Patients are stratified to one of two groups: Group 1 is patients on Gleevec or Tasigna who have been on drug less than 6 months; Group 2 is patients on Gleevec or Tasigna who have been on drug for equal to or more than 6 months.
  Group 1 is then divided into 2 groups: one using eMedonline for 3 months and the other not using eMedonline for 3 months. A crossover survey and pill counts will be done at the 3 month timepoint and then the groups will switch their access status to eMedonline.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wehbie, MD, Principal Investigator — Rex Cancer Center - Wakefield
Locations (3):
- United States (3):
  - UNC Healthcare, Chapel Hill, North Carolina
  - Rex Cancer Center, Raleigh, North Carolina
  - Rex Cancer Center - Wakefield, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No